CLINICAL TRIAL: NCT03706365
Title: A Phase 2/3, Randomized, Double-Blind, Placebo-Controlled Study of Abiraterone Acetate Plus Prednisone With or Without Abemaciclib in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of Abiraterone Acetate Plus Prednisone With or Without Abemaciclib (LY2835219) in Participants With Prostate Cancer
Acronym: CYCLONE 2
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16598; I3Y-MC-JPCM (Other: Eli Lilly and Company); 2016-004276-21 (EudraCT Number); 2023-506777-36-00 (EU CTIS Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2018-09-18; First posted 2018-10-16 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Metastatic Castration Resistant Prostate Cancer; mCRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abemaciclib; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abemaciclib (Experimental): Participants received 200 milligrams (mg) abemaciclib twice daily (BID) in combination with standard doses of 1000 mg abiraterone acetate once daily and 5 mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
  Interventions: Drug: Abemaciclib; Drug: Abiraterone acetate; Drug: Prednisone
- Placebo (Placebo Comparator): Participants received placebo BID in combination with standard doses of 1000 mg abiraterone acetate once daily and 5 mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
  Interventions: Drug: Placebo; Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abemaciclib — Administered orally.
  Other Names: LY2835219
  Arms: Abemaciclib
Drug: Placebo — Administered orally.
  Arms: Placebo
Drug: Abiraterone acetate — Administered orally.
Drug: Prednisone — Administered orally.

SUMMARY:
This study is being done to see how safe and effective abemaciclib is when given together with abiraterone acetate plus prednisone in participants with metastatic castration resistant prostate cancer. Prednisolone may be used instead of prednisone per local regulation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* Metastatic prostate cancer documented by positive bone scan and/or measurable soft tissue metastatic lesions by CT or magnetic resonance imaging (MRI).
* Progressive disease at study entry demonstrated during continuous androgen-deprivation therapy (ADT)/post orchiectomy defined as one or more of the following:

  * PSA progression
  * Radiographic progression per Response Evaluation Criteria in Solid Tumors (RECIST)1.1 for soft tissue and/or per Prostate Cancer Working Group 3 (PCWG3) for bone, with or without PSA progression
* Have adequate organ function.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.

Exclusion Criteria:

* Prior therapy with cytochrome P450 (CYP)17 inhibitors.
* Prior treatment with abemaciclib or any cyclin-dependent kinase (CDK) 4 & 6 inhibitors.
* Prior cytotoxic chemotherapy for metastatic castration resistant prostate cancer (participants treated with docetaxel in the metastatic hormone-sensitive prostate cancer [mHSPC] are eligible). Prior radiopharmaceuticals for prostate cancer, or prior enzalutamide, apalutamide, darolutamide or sipuleucel-T. Participants who had prior radiation or surgery to all target lesions.
* Currently enrolled in a clinical study involving an investigational product.
* Gastrointestinal disorder affecting the absorption or ability to swallow large pills.
* Clinically significant heart disease, active or chronic liver disease, moderate/severe hepatic impairment (Child-Pugh Class B and C).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (112):
- United States (33):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic in Arizona - Phoenix, Phoenix, Arizona
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - CBCC Global Research, Inc., Bakersfield, California
  - Providence St. Jude Medical Center, Fullerton, California
  - Moores Cancer Center, La Jolla, California
  - TRIO-US (Translational Research in Oncology-US), Los Angeles, California
  - UCLA Hematology/Oncology - Westwood (Building 100), Los Angeles, California
  - Pacific Cancer Care, Monterey, California
  - Sansum Clinic_Kendle, Santa Barbara, California
  - Rocky Mountain Cancer Center, Lone Tree, Colorado
  - Millennium Oncology - Hollywood, Hollywood, Florida
  - Northside Hospital, Atlanta, Georgia
  - Fort Wayne Medical Oncology And Hematology at Parkview Comprehensive Cancer Center, Fort Wayne, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - M Health Fairview University of Minnesota Medical Center - East Bank, Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology (NYOH) - Clifton Park Cancer Center, Albany, New York
  - Associated Medical Professionals - Urology, Syracuse, New York
  - Research Medical Center, Nashville, Tennessee
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - New York Oncology Hematology (NYOH) - Clifton Park Cancer Center, The Woodlands, Texas
  - Northwest Cancer Specialists PC, The Woodlands, Texas
  - Sansum Clinic_Kendle, The Woodlands, Texas
  - Texas Oncology - Longview Cancer Center, The Woodlands, Texas
  - Texas Oncology Cancer Care and Research Center, The Woodlands, Texas
  - Texas Oncology Fort Worth, The Woodlands, Texas
  - Texas Oncology-Memorial City, The Woodlands, Texas
  - US Oncology, The Woodlands, Texas
  - USO-Cancer Care Center of Brevard, Inc., The Woodlands, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - The University of Vermont Medical Center Inc., Burlington, Vermont
- Australia (6):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Southside Cancer Care Centre, Kogarah, New South Wales
  - Macquarie University, Macquarie University, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
- China (26):
  - Second Affiliated hospital of Anhui Medical University, Hefei, Anhui
  - Wannan Medical College Yijishan Hospital, Wuhu, Anhui
  - Lanzhou university second hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Centre, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical SchoolNanjing, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated Fudan University, Shanghai, Shanghai Municipality
  - Nanchong Central Hospital, Nanchong, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
- Denmark (2):
  - Rigshospitalet, Copenhagen, Capital Region
  - Næstved Sygehus, Næstved, Region Sjælland
- France (6):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Centre de Cancérologie du Grand Montpellier, Montpellier, Languedoc-Roussillon
  - Clinique Victor Hugo Le Mans, Le Mans, Pays de la Loire Region
  - CHD Vendee, La Roche-sur-Yon, Vendée
  - CHU de Bordeaux Hop St ANDRE, Bordeaux
  - Henri Mondor Hospital, Créteil, Île-de-France Region
- Germany (9):
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Gesundheitszentrum Holzminden, Holzminden, Lower Saxony
  - Studienzentrum Bayenthal Urologische Partnerschaft Köln, Cologne, North Rhine-Westphalia
  - Urologie Neandertal - Praxis Mettmann, Mettmann, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - Private Practice - Dr. Stammel & Dr. Garcia, Wesel, North Rhine-Westphalia
  - Private Practice - Dr. Silvio Szymula, Leipzig, Saxony
  - Private Practice - Dr. Ralf Eckert, Eisleben Lutherstadt, Saxony-Anhalt
- Japan (13):
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Saitama Prefectural Cancer Center, Ina-machi, Saitama
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Showa University Hospital, Shinagawa, Tokyo
  - Gifu University Hospital, Gifu
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Osaka International Cancer Institute, Osaka
- Netherlands (3):
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - St. Antonius Ziekenhuis, locatie Utrecht, Utrecht
- Romania (3):
  - Ovidius Clinical Hospital OCH, Ovidiu, Constanța County
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Gral Medical Diagnostic Center, Bucharest
- South Korea (4):
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Songpagu, Seoul-teukbyeolsi [Seoul]
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, Hospitalet, Barcelona [Barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital General Universitario Gregorio Marañon, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Smith M, Piulats J, Todenhofer T, Lee JL, Arija JA, Mazilu L, Azad A, Alonso-Gordoa T, McGovern U, Choudhury A, Horvath L, Ye D, Han W, Suzuki H, Uemura H, McKay R, Ades S, Flechon A, Pieczonka C, Fernandes MS, Hulstijn M, Lithio A, Nacerddine K, Agarwal N; CYCLONE 2 investigators. Abemaciclib plus abiraterone in patients with metastatic castration-resistant prostate cancer (CYCLONE 2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2025 Nov;26(11):1489-1500. doi: 10.1016/S1470-2045(25)00475-9. PMID 41167216
- See also: A Study of Abiraterone Acetate Plus Prednisone With or Without Abemaciclib (LY2835219) in Participants With Prostate Cancer — https://trials.lillytrialguide.com/en-US/trial/3gu4aah7luigAwcweY4wWK

RESULTS

PARTICIPANT FLOW:
Groups:
- Abemaciclib: Participants received 200 milligram (mg) abemaciclib twice daily (BID) in combination with standard doses of 1000 mg abiraterone acetate once daily and 5mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
- Placebo: Participants received placebo BID in combination with standard doses of 1000 mg abiraterone once daily and 5 mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
Period: Overall Study
Arm/Group | Abemaciclib | Placebo
Started | 206 | 187
Received at Least One Dose of Study Drug | 206 | 185
Completed | 131 | 121
Not Completed | 75 | 66
Not completed — Lost to Follow-up | 7 | 0
Not completed — Withdrawal by Subject | 17 | 15
Not completed — On Study Treatment | 51 | 51

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Abemaciclib: Participants received 200 mg abemaciclib BID in combination with standard doses of 1000 mg abiraterone acetate once daily and 5mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
- Total: Total of all reporting groups
Arm/Group | Abemaciclib | Placebo | Total
Number analyzed (Participants) | 206 | 187 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.70 (8.57) | 69.60 (8.81) | 69.10 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 206 | 187 | 393
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 7 | 20
  Not Hispanic or Latino | 186 | 174 | 360
  Unknown or Not Reported | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 45 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 161 | 128 | 289
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  Australia | 17 | 18 | 35
  China | 4 | 9 | 13
  Denmark | 7 | 10 | 17
  France | 4 | 5 | 9
  Germany | 23 | 16 | 39
  Japan | 15 | 18 | 33
  Netherlands | 7 | 8 | 15
  Romania | 10 | 7 | 17
  South Korea | 14 | 17 | 31
  Spain | 45 | 30 | 75
  United Kingdom | 11 | 9 | 20
  United States | 49 | 40 | 89

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression Free Survival (rPFS)
Description: The rPFS time is measured from the date of randomization to the earliest date of investigator determined radiographic disease progression (by objective radiographic disease assessment per response evaluation criteria in solid tumors (RECIST) version 1.1 for soft tissue AND/OR radionuclide bone scan using prostate cancer working group 3 -PCWG3 criteria for bone) or death from any cause, whichever occurs first.
Time Frame: From Date of Randomization to Radiographic Disease Progression or Death from Any Cause (Up to 60 Months)
Population: All randomized participants. Participants were analyzed according to the treatment arm they were assigned to regardless of what actual treatment they received.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Abemaciclib: Participants received 200 mg abemaciclib BID in combination with standard doses of 1000 mg abiraterone acetate once daily and 5 mg prednisone BID administered orally on a continuous dosing schedule on days 1 through 28 of a 28-day cycle until radiographic and/or symptomatic progression or until another discontinuation criterion is met.
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 206 | 187
Months | 21.96 [19.33 to 27.48] | 20.28 [16.47 to 24.36]
Statistical Analysis 1: Comparison: Abemaciclib vs Placebo; Test type: Other; p = 0.2123, Log Rank; Hazard Ratio (HR) = 0.829, 95% CI 2-sided [0.619 to 1.111]

2. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: The PSA progression is defined as a greater than or equal to (>=) 25 percentage (%) increase and an absolute increase of >=2 nanogram/milliliter (ng/mL) above the nadir (or baseline value if baseline is the smallest on study), which is confirmed by a second value obtained 3 or more weeks later.
Time Frame: From Date of Randomization to the Date of the First Observation of PSA Progression (Up to 60 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 206 | 187
Months | 22.19 [15.68 to 33.17] | 16.60 [12.03 to 20.28]
Statistical Analysis 1: Comparison: Abemaciclib vs Placebo; Test type: Other; p = 0.0026, Log Rank; Hazard Ratio (HR) = 0.637, 95% CI 2-sided [0.474 to 0.856]

3. Secondary Outcome: Radiographic Progression Free Survival (rPFS) Determined by Blinded Independent Central Review
Description: rPFS is defined as the time from the date of randomization to the earliest date of radiographic disease progression determined by blinded independent central review (BICR) or death from any cause, whichever occurs first.
Time Frame: From Date of Randomization Until Radiographic Disease Progression or Death from Any Cause (Up to 60 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 206 | 187
Months | 24.89 [21.96 to NA] — Upper limit of 95% confidence interval was not achieved due to insufficient sample data. | 22.88 [19.36 to 31.50]
Statistical Analysis 1: Comparison: Abemaciclib vs Placebo; Test type: Other; p = 0.2899, Log Rank; Hazard Ratio (HR) = 0.842, 95% CI 2-sided [0.611 to 1.160]

4. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With a Complete Response (CR) or Partial Response (PR)
Description: ORR is a summary measure of best overall response (BOR) as defined by RECIST 1.1 for soft tissue per investigator assessment. BOR is derived from time point responses. All time point responses observed while on study treatment and during the short-term follow-up period (but before the initiation of post-discontinuation systemic anticancer therapy) will be included in the derivation.
  Each patient's BOR will be categorized as complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or not evaluable (NE). A BOR of CR or PR will require confirmation, but sensitivity analyses of response-based endpoints may be performed where confirmation of a BOR of CR or PR is not required.
Time Frame: Baseline to Radiographic Disease Progression (Up to 60 Months)
Population: All randomized participants who received at least one dose of the study drug and had CR or PR responses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 84 | 73
percentage of participants | 45.2 [34.6 to 55.9] | 54.8 [43.4 to 66.2]

5. Secondary Outcome: Duration of Response (DOR)
Description: The DoR time is defined only for responders (participants with a soft tissue BOR of CR or PR) in the measurable disease population. It is measured from the date of first evidence of soft tissue CR or PR to the earliest date of investigator determined radiographic disease progression or death from any cause, whichever is earlier.
Time Frame: Date of First Documented CR or PR to Date of Radiographic Disease Progression or Death from Any Cause (Up to 60 Months)
Population: All randomized participants who received at least one dose of the study drug and had CR or PR responses with objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 38 | 40
Months | 21.27 [16.60 to NA] — Upper limit of 95% confidence interval was not achieved due to insufficient sample data. | 15.68 [11.87 to 39.35]
Statistical Analysis 1: Comparison: Abemaciclib vs Placebo; Test type: Other; p = 0.3531, Log Rank; Hazard Ratio (HR) = 0.731, 95% CI 2-sided [0.377 to 1.419]

6. Secondary Outcome: Overall Survival (OS)
Description: The OS time is measured from the date of randomization to the date of death from any cause. If the participant was alive or lost to follow-up at the time of data analysis, OS data were censored on the last date the participant was known to be alive.
Time Frame: From Date of Randomization to Date of Death Due to Any Cause (Up to 60 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 206 | 187
Months | 38.01 [30.58 to 46.65] | 33.21 [29.52 to NA] — Upper limit of 95% confidence interval was not achieved due to insufficient sample data.
Statistical Analysis 1: Comparison: Abemaciclib vs Placebo; Test type: Other; p = 0.6507, Log Rank; Hazard Ratio (HR) = 0.927, 95% CI 2-sided [0.669 to 1.285]

7. Secondary Outcome: Time to Symptomatic Progression
Description: Time to symptomatic progression is defined as the time from randomization to any of the following (whichever occurs earlier):
  1. Symptomatic Skeletal Event (SSE), defined as symptomatic fracture, surgery or radiation to bone, or spinal cord compression.
  2. Pain progression or worsening of disease-related symptoms requiring initiation of a new systemic anti-cancer therapy.
  3. Development of clinically significant symptoms due to loco-regional tumor progression requiring surgical intervention or radiation therapy.
Time Frame: From Randomization to the Date of the First Documented Symptomatic Progression (Up to 60 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 206 | 187
Months | 51.39 [27.98 to NA] — Upper limit of 95% confidence interval was not achieved due to high censoring rate. | 35.74 [28.44 to NA] — Upper limit of 95% confidence interval was not achieved due to high censoring rate.
Statistical Analysis 1: Comparison: Abemaciclib vs Placebo; Test type: Other; p = 0.1807, Log Rank; Hazard Ratio (HR) = 0.768, 95% CI 2-sided [0.522 to 1.131]

8. Secondary Outcome: Pharmacokinetics (PK): Mean Steady State Exposure of Abemaciclib
Description: PK: Mean steady state exposure of abemaciclib.
Time Frame: Cycle (C) 1 Day (D) 1: Predose, 30 min post-dose; C1 D15, C2 D1, C2 D15, C3 D1: Post dose (28 Days Cycle)
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Abemaciclib
Number analyzed (Participants) | 170
nanogram per milliliter (ng/mL)
  C1 D1: number analyzed (Participants) | 79
  C1 D1 | 4.79 (157)
  C1 D15: number analyzed (Participants) | 141
  C1 D15 | 289 (58.7)
  C2 D1: number analyzed (Participants) | 117
  C2 D1 | 253 (65.7)
  C2 D15: number analyzed (Participants) | 95
  C2 D15 | 252 (68.4)
  C3 D1: number analyzed (Participants) | 81
  C3 D1 | 270 (54.5)

9. Secondary Outcome: PK: Mean Steady State Exposure of Abemaciclib Metabolite LSN2839567
Description: PK: Mean steady state exposure of abemaciclib metabolite LSN2839567.
Time Frame: C1 D1: Predose, 30 min post-dose; C1 D15, C2 D1, C2 D15, C3 D1: Post dose (28 Days Cycle)
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Abemaciclib
Number analyzed (Participants) | 170
ng/mL
  C1 D1: number analyzed (Participants) | 65
  C1 D1 | 2.90 (87.4)
  C1 D15: number analyzed (Participants) | 137
  C1 D15 | 125 (50.4)
  C2 D1: number analyzed (Participants) | 115
  C2 D1 | 112 (50.1)
  C2 D15: number analyzed (Participants) | 94
  C2 D15 | 116 (51.0)
  C3 D1: number analyzed (Participants) | 81
  C3 D1 | 110 (62.2)

10. Secondary Outcome: PK: Mean Steady State Exposure of Abemaciclib Metabolite LSN3106726
Description: PK: Mean steady state exposure of abemaciclib metabolite LSN3106726.
Time Frame: C1 D1: Predose, 30 min post-dose; C1 D15, C2 D1, C2 D15, C3 D1: Post dose (28 Days Cycle)
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Abemaciclib
Number analyzed (Participants) | 170
ng/mL
  C1 D1: number analyzed (Participants) | 59
  C1 D1 | 2.80 (77.7)
  C1 D15: number analyzed (Participants) | 137
  C1 D15 | 195 (43.0)
  C2 D1: number analyzed (Participants) | 115
  C2 D1 | 174 (42.8)
  C2 D15: number analyzed (Participants) | 94
  C2 D15 | 174 (44.1)
  C3 D1: number analyzed (Participants) | 80
  C3 D1 | 176 (36.4)

11. Secondary Outcome: PK: Mean Steady State Exposure of Abiraterone Acetate
Description: PK: Mean Steady State Exposure of Abiraterone Acetate.
Time Frame: C1 D15, Post dose
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 189 | 175
ng/mL | 45.2 (175) | 40.0 (203)

12. Secondary Outcome: Time to Worst Pain Progression
Description: Time to Worst Pain Progression defined as the time from randomization to any of the following (whichever occurs earlier): For participants without opioid use at baseline (World Health Organization-Analgesic Ladder-WHO-AL ≤ 2):- Worst pain progression (an increase of 2 points from baseline on the Worst Pain Numeric Rating Scale (NRS) item on 2 consecutive evaluations), Initiation of weak or strong opioids (WHO-AL ≥ 3); For participants with weak or strong opioid use at baseline (WHO-AL ≥ 3): Worst pain progression (an increase of 2 points from baseline on the Worst Pain NRS item on 2 consecutive evaluations) without concurrent decreased opioid use (a decrease in WHO-AL of 1 or more) -Increased opioid use (an increase in WHO-AL of 1 or more).
Time Frame: From Randomization Through Follow-up (Up to 60 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Placebo
Number analyzed (Participants) | 206 | 187
Months | 41.49 [19.40 to NA] — Upper limit of 95% confidence interval was not achieved due to insufficient sample data. | 24.79 [19.17 to 31.46]
Statistical Analysis 1: Comparison: Abemaciclib vs Placebo; Test type: Other; p = 0.6970, Log Rank; Hazard Ratio (HR) = 0.935, 95% CI 2-sided [0.665 to 1.314]

ADVERSE EVENTS:
Time Frame: Baseline Up to 60 Months
Description: All-Cause Mortality: All randomized participants. Serious and other adverse events: All participants who received at least one dose of the study drug, regardless of their eligibility for the study.
Arm/Group | Abemaciclib | Placebo
All-Cause Mortality (participants affected / at risk) | 81/206 | 72/187
Serious Adverse Events (participants affected / at risk) | 89/206 | 66/185
Other Adverse Events (participants affected / at risk) | 204/206 | 176/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=206) | Placebo (N=185)
Anaemia (Blood and lymphatic system disorders) | 6 (8) | 3 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (3)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Anal abscess (Infections and infestations) | 1 (2) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Covid-19 (Infections and infestations) | 4 (5) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Device related bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (7) | 5 (5)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (4) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (2)
Urosepsis (Infections and infestations) | 4 (5) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Colloid brain cyst (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (2)
Spinal cord compression (Nervous system disorders) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 9 (9) | 1 (1)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 3 (4)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Embolism arterial (Vascular disorders) | 1 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=206) | Placebo (N=185)
Anaemia (Blood and lymphatic system disorders) | 91 (164) | 21 (30)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (6)
Leukopenia (Blood and lymphatic system disorders) | 39 (78) | 3 (3)
Lymph node pain (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 19 (24) | 13 (26)
Neutropenia (Blood and lymphatic system disorders) | 57 (135) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 34 (56) | 5 (6)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 4 (5) | 3 (5)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Atrial flutter (Cardiac disorders) | 3 (3) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (4)
Cardiac septal hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 4 (4) | 4 (4)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 6 (6)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 1 (2)
Tachycardia (Cardiac disorders) | 7 (7) | 3 (4)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 3 (3)
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 3 (4)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 1 (1)
Cushingoid (Endocrine disorders) | 4 (4) | 5 (5)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Pituitary-dependent cushing's syndrome (Endocrine disorders) | 2 (2) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 6 (6) | 4 (7)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Corneal erosion (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 5 (5) | 0 (0)
Episcleritis (Eye disorders) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 1 (2) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 1 (2) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 1 (1)
Lacrimation increased (Eye disorders) | 14 (18) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 2 (2) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 5 (6) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 39 (53) | 25 (30)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 41 (57) | 35 (43)
Dental caries (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dental pulp disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 134 (414) | 35 (76)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 10 (12) | 5 (5)
Duodenal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 23 (27) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 6 (7) | 4 (4)
Food poisoning (Gastrointestinal disorders) | 1 (4) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (11) | 7 (7)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 12 (12) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 4 (4) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 1 (1)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 73 (121) | 27 (32)
Odynophagia (Gastrointestinal disorders) | 4 (5) | 1 (1)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral mucosa haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Peritoneal lesion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 5 (5) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 5 (6) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 10 (12) | 2 (2)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 5 (5)
Vomiting (Gastrointestinal disorders) | 48 (63) | 17 (31)
Axillary pain (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 4 (4) | 0 (0)
Chest pain (General disorders) | 2 (2) | 4 (5)
Chills (General disorders) | 6 (7) | 3 (3)
Crying (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 2 (2) | 3 (3)
Fatigue (General disorders) | 107 (196) | 47 (74)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 2 (2) | 0 (0)
Inflammatory pain (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 7 (8) | 4 (5)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 2 (2)
Localised oedema (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 5 (6) | 4 (4)
Mucosal inflammation (General disorders) | 5 (8) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 2 (2)
Oedema (General disorders) | 1 (1) | 5 (8)
Oedema peripheral (General disorders) | 41 (61) | 23 (29)
Pain (General disorders) | 7 (7) | 2 (2)
Peripheral swelling (General disorders) | 5 (6) | 0 (0)
Physical deconditioning (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 21 (33) | 14 (17)
Swelling (General disorders) | 0 (0) | 1 (1)
Swelling face (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (3) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 5 (10) | 0 (0)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Balanitis candida (Infections and infestations) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Candida infection (Infections and infestations) | 2 (3) | 0 (0)
Cellulitis (Infections and infestations) | 4 (6) | 2 (2)
Conjunctivitis (Infections and infestations) | 5 (8) | 2 (3)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 32 (39) | 28 (28)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 2 (2)
Fungal tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 7 (7) | 4 (4)
Gingivitis (Infections and infestations) | 2 (2) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3)
Hordeolum (Infections and infestations) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 5 (5)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (8) | 5 (7)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal infection (Infections and infestations) | 1 (1) | 1 (1)
Onychomycosis (Infections and infestations) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 3 (3) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 2 (2)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 6 (6)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 1 (2) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 3 (3)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Syphilis (Infections and infestations) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 2 (2)
Tooth infection (Infections and infestations) | 4 (7) | 2 (2)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 7 (8)
Urinary tract infection (Infections and infestations) | 15 (21) | 21 (33)
Viral infection (Infections and infestations) | 4 (4) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Wound infection (Infections and infestations) | 3 (3) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (4)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 14 (14) | 10 (11)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 26 (36) | 13 (24)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ocular procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 9 (10) | 4 (5)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (6) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase decreased (Investigations) | 0 (0) | 1 (3)
Alanine aminotransferase increased (Investigations) | 48 (68) | 21 (40)
Alpha 1 microglobulin increased (Investigations) | 0 (0) | 1 (4)
Amylase increased (Investigations) | 1 (2) | 1 (1)
Apolipoprotein a-i increased (Investigations) | 0 (0) | 1 (1)
Apolipoprotein b decreased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase decreased (Investigations) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 36 (43) | 15 (19)
Bile acids increased (Investigations) | 1 (4) | 0 (0)
Bleeding time prolonged (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 10 (16) | 8 (11)
Blood bilirubin decreased (Investigations) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 5 (10) | 2 (5)
Blood cholesterol decreased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase decreased (Investigations) | 0 (0) | 1 (3)
Blood creatine phosphokinase increased (Investigations) | 6 (6) | 2 (2)
Blood creatinine decreased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 58 (126) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 3 (4) | 7 (7)
Blood urea increased (Investigations) | 7 (7) | 2 (6)
Blood uric acid increased (Investigations) | 1 (3) | 0 (0)
Bone scan abnormal (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (2)
Cardiac ventriculogram left abnormal (Investigations) | 1 (1) | 0 (0)
Complement factor c1 decreased (Investigations) | 0 (0) | 1 (3)
Cystatin c increased (Investigations) | 4 (4) | 1 (3)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1)
Electrocardiogram st-t segment abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram u-wave abnormality (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 5 (10) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 3 (9) | 1 (1)
Glomerular filtration rate increased (Investigations) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 3 (3) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Monocyte count increased (Investigations) | 0 (0) | 2 (6)
Muscle strength abnormal (Investigations) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 2 (4)
Nitrite urine present (Investigations) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 1 (1) | 0 (0)
Sars-cov-2 test positive (Investigations) | 4 (4) | 0 (0)
Serum ferritin decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (4) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 1 (1)
Vitamin b12 decreased (Investigations) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 23 (31) | 10 (11)
Weight increased (Investigations) | 3 (4) | 6 (7)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 50 (70) | 15 (17)
Dehydration (Metabolism and nutrition disorders) | 8 (10) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Food aversion (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 1 (5)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 (11) | 5 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (19) | 14 (19)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (8)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (9) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 16 (24) | 7 (11)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (3) | 2 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (8) | 5 (11)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (37) | 13 (20)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (12) | 5 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 14 (17) | 4 (8)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 (49) | 34 (45)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (44) | 42 (57)
Bone loss (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 12 (14)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (7)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 (15) | 21 (24)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 (13) | 10 (10)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 15 (22) | 12 (16)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (8)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (15) | 10 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 7 (7)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (3)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 (24) | 17 (21)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1)
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 2 (2) | 3 (3)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 3 (3) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 29 (35) | 15 (17)
Dizziness postural (Nervous system disorders) | 3 (3) | 2 (2)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 25 (29) | 4 (4)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspraxia (Nervous system disorders) | 1 (1) | 0 (0)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 16 (21) | 16 (22)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 3 (3) | 2 (2)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 3 (3) | 3 (4)
Meralgia paraesthetica (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Muscle spasticity (Nervous system disorders) | 1 (2) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy (Nervous system disorders) | 18 (20) | 14 (14)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Primary stabbing headache (Nervous system disorders) | 0 (0) | 1 (2)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 2 (2) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 6 (8) | 3 (3)
Taste disorder (Nervous system disorders) | 6 (8) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 6 (7) | 1 (1)
Vascular parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (6) | 4 (4)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
Bruxism (Psychiatric disorders) | 2 (2) | 0 (0)
Claustrophobia (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 10 (11) | 3 (3)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (2)
Dissociation (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 19 (20) | 15 (17)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 3 (3) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 6 (7) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder hypertrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 13 (16) | 7 (8)
Glycosuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 21 (25) | 17 (28)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 2 (6)
Micturition urgency (Renal and urinary disorders) | 4 (4) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (5) | 0 (0)
Nocturia (Renal and urinary disorders) | 11 (13) | 10 (10)
Pollakiuria (Renal and urinary disorders) | 9 (9) | 14 (15)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (11) | 2 (2)
Renal colic (Renal and urinary disorders) | 2 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (5) | 1 (1)
Renal impairment (Renal and urinary disorders) | 6 (6) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 2 (2)
Sterile pyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteral disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 7 (7)
Urinary retention (Renal and urinary disorders) | 2 (2) | 5 (7)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 5 (6) | 6 (7)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prostatic disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Retracted nipple (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 45 (59) | 20 (22)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (31) | 15 (16)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperactive pharyngeal reflex (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (5)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Pulmonary artery dilatation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (18) | 4 (4)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (9) | 3 (3)
Angiodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (11) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 6 (9) | 2 (2)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Koilonychia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 13 (13) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (12) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 21 (28) | 11 (11)
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sensitive skin (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Skin atrophy (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin dystrophy (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin fragility (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 7 (8) | 4 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Symmetrical drug-related intertriginous and flexural exanthema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Capillary fragility (Vascular disorders) | 5 (5) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 5 (6) | 1 (1)
Haematoma (Vascular disorders) | 5 (5) | 3 (3)
Hot flush (Vascular disorders) | 25 (27) | 24 (27)
Hypertension (Vascular disorders) | 24 (36) | 34 (63)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 9 (9) | 3 (3)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 2 (2) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 2 (2) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Vascular fragility (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT03706365/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT03706365/SAP_001.pdf